CLINICAL TRIAL: NCT07073820
Title: A PHASE 2, OPEN-LABEL EXTENSION STUDY TO INVESTIGATE THE SAFETY AND EFFICACY OF PF-07868489 ADMINISTERED TO ADULT PARTICIPANTS WITH PULMONARY ARTERIAL HYPERTENSION
Brief Title: A Study to Learn About the Study Medicine (Called PF-07868489) in People With Pulmonary Arterial Hypertension Who Have Previously Participated in a Clinical Study With PF-07868489
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C5001004; 2025-521155-23-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Open Label (Experimental): Participants will receive subcutaneous doses of PF-07868489 every 4 weeks
  Interventions: Drug: PF-07868489

INTERVENTIONS:
Drug: PF-07868489 — Participants will receive subcutaneous doses of PF-07868489 every 4 weeks

SUMMARY:
The purpose of this study is to learn about the long-term safety, tolerability and effects of the study medicine (PF-07868489) for the possible treatment of PAH. PAH is a condition in which there is high blood pressure in the arteries that carry blood from the heart to the lungs. This high pressure makes it harder for the heart to pump blood through those lungs, potentially damaging the right side of the heart.

This is an open-label study. Which means that both the healthcare providers and the study participants are aware of the medicine being given. This study is also an extension study with study medicine (PF-07868489). An extension study allows patients from an earlier clinical study (also called as qualifying study) to continue participating to assess long-term benefits and safety of the medicine.

ELIGIBILITY:
This study is seeking participants who are:

* aged 18 years or older at screening of the previous study and completed the required treatment duration with PF-07868469 and other assessments at the end of that study.
* willing and able to abide with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
* do not have worsening or hospitalization for worsening PAH during the qualifying study.
* not on placement for a surgery to replace any tissue or part of the body (transplant), and planned surgery for PAH.
* do not have an ongoing major health issue in the qualifying study, which in the opinion of the study doctor could make the participant not qualify for this study.
* not suffering from or in the past have suffered from hepato-pulmonary syndrome (liver-related lung problem).
* not currently prescribed or taking medicines called as GLP-1 agonist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2029-01-08 (Estimated); Study Completion 2029-01-08 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) | Baseline up to week 111
Number of Participants With Change From Baseline in Laboratory Tests Results | Baseline up to week 111
Number of Participants With Vital Sign Abnormalities | Baseline up to week 111

SECONDARY OUTCOMES:
Number of Participants With Change From Baseline in Electrocardiogram (ECG) Parameters | Baseline up to week 111
Change From Baseline in N-Terminal Prohormone Brain Natriuretic Peptide (NT-proBNP) Concentration | Baseline up to week 104
Minimum Observed Plasma Trough Concentration (Cmin), as data permits | Baseline up to week 111
Incidence of Anti-Drug Antibody (ADA) | Baseline up to week 111

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (26):
- United States (5):
  - UCSF Health St. Mary's Hospital, San Francisco, California
  - Heart and Vascular Center, San Francisco, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Norton Hospital, Louisville, Kentucky
  - Norton Pulmonary Specialists, Louisville, Kentucky
- Royal Prince Alfred Hospital, Camperdown, New South Wales, Australia
- Canada (2):
  - London Health Sciences Centre - University Hospital, London, Ontario
  - London Health Sciences Centre, London, Ontario
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China
- Germany (5):
  - Thoraxklinik-Heidelberg gGmbH, Heidelberg, Baden-Wurttemberg
  - Universitätsklinikum Regensburg, Regensburg, Bavaria
  - Universitaetsklinikum Giessen und Marburg GmbH, Giessen, Hesse
  - Universitätsmedizin Greifswald, Greifswald, Mecklenburg-Vorpommern
  - Universitaetsklinikum Carl Gustav Carus, Technischen Universitaet Dresden, Dresden, Saxony
- Japan (4):
  - Kobe University Hospital, Kobe, Hyōgo
  - St. Marianna University Hospital, Kawasaki, Kanagawa
  - Tohoku University Hospital, Sendai, Miyagi
  - National Hospital Organization Okayama Medical Center, Okayama
- South Korea (4):
  - Gachon University Gil Medical Center, Incheon, Incheon-gwangyeoksi [incheon]
  - Seoul National University Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul-teukbyeolsi [seoul]
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [seoul]
- Spain (3):
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitario La Paz, Madrid, Madrid, Comunidad de
  - Hospital Universitario 12 de Octubre, Madrid
- Hammersmith Hospital, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5001004